CLINICAL TRIAL: NCT05710016
Title: Evaluation Of Intra-Operative Neuro-Monitoring Alarm During Complex Spine Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, shady nady zaky, principle investigator, Assiut University
Other Study IDs: Spine Surgery Neuromonitoring
Record Dates: First submitted 2023-01-25; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Spine Injuries and Disorders
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Iatrogenic spinal cord injury is the most feared complication of complex spine surgery. The incidence of neurological complications for spinal deformity surgery has been estimated by the Scoliosis Research Society as 1%, except when a combined approach is used, where the rate increases to 1.87% [1]. Intraoperative neuromonitoring (IONM) techniques are usually implemented during spine surgery to avoid nefarious abuse of the nervous system, which can cause postoperative problem [2].

In 1992 a Scoliosis Research Society study concluded that the use of intraoperative spinal cord neurophysiological monitoring during operative procedures including instrumentation should be considered ''a viable alternative as well as an adjunct to the use of the wake-up test during spinal surgery'' [5]. The benefit of using neuromonitoring has been validated by numerous studies involving scoliosis correction, revision surgeries and vertebral osteotomies.

DETAILED DESCRIPTION:
The trend in IONM usage in the current literature, which may be a direct consequence of improved efficacy of the procedure, and the development of optimized treatment algorithm [6]. Nevertheless, it is well known that the use of somatosensory evoked potentials (SEPs) alone may be ineffective in detecting a motor tract deficit [7, 8]. As a result, various methods for monitoring the motor tract of the spinal cord have been developed. The most commonly used stimulation technique is transcranial electric stimulation (TES) of the primary motor cortex by corkscrew electrodes placed in the scalp, to produce myogenic motor evoked potential[9]. The combination of SEPs and TES-MEPs provides global monitoring coverage of spinal cord function [10]. Based on the available evidence, it is recommended that the use of multimodality neuromonitoring be considered in complex spine surgery where the spinal cord or nerve roots are deemed to be at risk [11].

ELIGIBILITY:
Inclusion Criteria:

* patient with spine deformities
* patient with sever cervical and lumbar degenerative diseases
* patient with combined cervical and lumbar diseases
* patient with spine tumours

Exclusion Criteria:

• cases with mild to moderate degenerative diseases simple spine procedures

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All cases arrived in our facility meets our inclusion criteria within one year .
  Estimated number of cases based on our hospital records for the last year was 64 cases .
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Measurement the incidence of new neurologic deficits (NNDs) and estimate sensitivity and specificity of IONM modalities | immediate measurement
  neurological examination